CLINICAL TRIAL: NCT00285324
Title: Two-Compartment Model of Diffusion Tensor Magnetic Resonance Imaging (DT-MRI) for the Diagnosis of Glioma Tumor Recurrence Versus Radiation Necrosis
Brief Title: Diffusion Tensor MRI to Distinguish Brain Tumor Recurrence From Radiation Necrosis
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060085; 06-N-0085
Record Dates: First submitted 2006-02-01; First posted 2006-02-01 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-08-20

CONDITIONS: Glioma Tumor Recurrence; Radiation Necrosis; Primary Brain Tumor
Keywords: Glioma; Glioblastoma Multiforme; Brain Cancer; Diffusion-Weighted Magnetic Resonance Imaging; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Glioma; Glioblastoma

SUMMARY:
This study will examine the use of a variation of standard magnetic resonance imaging (MRI) called diffusion tensor MRI (DT-MRI) for distinguishing injured brain tissue due to radiation therapy (radiation necrosis) from the return of a brain tumor that was previously removed (tumor recurrence). DT-MRI differs from standard MRI in the way that computers process the images; there is no difference in the experience of having the procedure done. Both radiation necrosis and tumor recurrence can occur within weeks to months following brain radiation treatment. Because the treatment and management options for the two conditions differ significantly, distinguishing the two is of critical importance. Currently, surgical biopsy is required to make this differentiation.

Healthy volunteers and patients who have received radiation therapy as part of their treatment for a brain tumor may be eligible for this study. All candidates must be at least 21 years old. Patients must have a new area of abnormality that requires a biopsy to determine whether it is a tumor recurrence or radiation necrosis. Candidates are screened with a medical history and physical examination. In addition, patients have blood and urine tests.

All participants undergo MRI and DT-MRI. MRI uses a strong magnetic field and radio waves instead of X-rays to obtain images of body organs and tissues. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, the subject lies on a table that can slide in and out of the cylinder and wears earplugs to muffle loud knocking noises that occur during the scanning. Scanning time varies from 20 minutes to 3 hours, with most scans lasting 40-60 minutes. Subjects may be asked to lie still for up to 20 minutes at a time. DT-MRI is a type of MRI that measures how water moves in the brain tissue. This technique uses the same MRI machine as conventional MRI, but the diffusion images are obtained after the normal MRI scan, and by a computer program that is installed into the machine. This completes the participation of healthy subjects.

In addition to the scans, patients undergo brain biopsy of the abnormal areas identified by MRI. Patients' commitment to the study protocol is fulfilled when the surgery is complete; they may, however, continue to receive follow-up care at the NIH Clinical Center after they complete the study. They are given the results of the biopsy so that further treatment, if necessary, can be arranged.

DETAILED DESCRIPTION:
The most common major side effect of radiation therapy for the treatment of primary brain tumors is the necrosis of normal brain tissues (radiation necrosis). Radiation necrosis typically occurs weeks to months following treatment. The diagnosis is suspected when patients have new areas of gadolinium enhancement on magnetic resonance imaging (MRI) scans. Tumor recurrence can also occur within weeks to months following treatment and is represented by new areas of gadolinium enhancement as well. As the management options for radiation necrosis and tumor recurrence are significantly different, distinguishing the two is of critical importance. Conventional MRI, diffusion-weighted MRI (DW-MRI), MR spectroscopy, SPECT, and PET imaging have all been used to try to make this distinction, but the sensitivity and specificity of these techniques have not been clinically useful. Most patients must therefore undergo a risky diagnostic surgical procedure. Diffusion tensor MRI (DT-MRI) is an imaging technique that provides information regarding both the diffusive properties of water as well as the directionality of water movement. A modification of DT-MRI, referred to as two-compartment DT-MRI, appears to be more sensitive than other variations of MRI for the diagnosis of selected types of brain abnormalities.

Objective: We plan to conduct a feasibility study to determine if two-compartment DT-MRI can distinguish tumor recurrence from radiation necrosis.

Study Population: Patients aged greater than or equal to twenty one years old with a prior diagnosis of primary brain tumor and history of radiation treatment who develop new areas of gadolinium enhancement on conventional MRI scans and who require surgery for diagnostic or therapeutic purposes will be evaluated for enrollment in this study. Ten patient controls will also undergo DT-MRI scans for the purpose of obtaining normative data for this quantitative study.

Design: Patients who meet eligibility criteria will undergo a two compartment DT-MRI scan. Regions of abnormality will be identified and surgical biopsies will be obtained of these regions. The radiographic and histologic characteristics of the samples will be correlated. Volunteers will undergo DT-MRI scans only.

Outcome Measure: The primary outcome measure of this study is the degree of agreement between the radiographically predicted diagnosis of tumor recurrence or radiation necrosis using two-compartment DT-MRI and the histologic diagnosis of such. This outcome will be measured as the proportion of instances in which the two modalities identify a particular lesion as being tumor recurrence or as being radiation necrosis. The information gathered from this study will allow for the implementation of a larger study with more patients if there is a high degree of agreement between the two compartment DT-MRI and histologic diagnoses of surgical biopsy specimens. The long range goal of the larger study is to radiographically diagnose tumor recurrence or radiation necrosis with a high enough level of sensitivity and specificity to avoid a diagnostic surgical procedure with its attendant risks.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must:

Have a histologically confirmed glioma, for which radiation therapy has been previously administered.

Be able to undergo an MRI scan of the brain.

Have contrast enhancing lesions that are amendable to surgical biopsy and/or resection.

Be appropriate for an operative procedure as determined by a neurosurgeon and anesthesiologist.

Ten patient controls will be included in this study to foster technical development and for the acquisition of normative data. Patient controls will have defined unilateral abnormalities on previously obtained MRI scans, but will not have had radiation treatment.

Be greater than or equal to 21 years of age.

EXCLUSION CRITERIA:

Patients must not:

Have any of the following: aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker or auto defibrillator, cochlear implant, ocular foreign body or implant (e.g. metal shavings, retinal clips), or insulin pump as these items would be contra-indications to undergoing an MRI scan.

Be poor operative candidates from an anesthetic point of view secondary to other major medical illnesses - the risk of undergoing general anesthesia outweighs the potential benefit of the clinical information gained from a surgical biopsy/resection.

Have a coagulopathy demonstrated by an abnormal prothrombin time, activated partial thromboplastin time, or thrombocytopenia (platelet count less that 150,000 platelets/mm3) - the risk of developing uncontrollable intra-operative bleeding outweighs the potential benefit of the clinical information gained from a surgical biopsy/resection.

Significant psychiatric impairments which, in the opinion of the investigators, will interfere with the proper administration or completion of the protocol - self explanatory.

Acute or untreated infections (viral, bacterial or fungal) - patients with active infections are highly likely to have spread of their infections to the brain as a result of a biopsy/resection.

Be pregnant at the time of the treatment - Women who are pregnant or nursing are excluded from this protocol. Therefore, all women of childbearing potential will have a pregnancy test performed, which must be negative, before proceeding. General anesthesia and surgery may subject the fetus to unacceptable risks. Also, the NIH does not offer full obstetrical services in the event that medical care to the mother and/or fetus is required.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01-27; Study Completion 2013-08-20

CONTACTS AND LOCATIONS:
Overall Officials: John K Park, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ammirati M, Galicich JH, Arbit E, Liao Y. Reoperation in the treatment of recurrent intracranial malignant gliomas. Neurosurgery. 1987 Nov;21(5):607-14. doi: 10.1227/00006123-198711000-00001. PMID 2827051
- [Background] Basser PJ, Mattiello J, LeBihan D. MR diffusion tensor spectroscopy and imaging. Biophys J. 1994 Jan;66(1):259-67. doi: 10.1016/S0006-3495(94)80775-1. PMID 8130344
- [Background] Biousse V, Newman NJ, Hunter SB, Hudgins PA. Diffusion weighted imaging in radiation necrosis. J Neurol Neurosurg Psychiatry. 2003 Mar;74(3):382-4. doi: 10.1136/jnnp.74.3.382. PMID 12588935